CLINICAL TRIAL: NCT03561766
Title: Birth Cohort Study of China Medical University in Shenyang
Brief Title: Birth Cohort Study of China Medical University
Status: Recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caixia Liu, Director of the second obstetrical department, Shengjing Hospital
Other Study IDs: CMUBCS
Record Dates: First submitted 2018-05-21; First posted 2018-06-19 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Twin; Complicating Pregnancy; Advanced Maternal Age Pregnancy; Scarred Uterus; Overweight and Obesity
MeSH Terms: conditions — Pregnancy Complications; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During pregnancy: maternal blood, urine and stool ; fetal blood and oral mucosal cell At delivery: cord, cord blood and placenta During Infancy：dry blood spot During childhood: blood, buccal swab and stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The CMUBCS is a birth cohort study located in Shenyang, China. Its initial aim is to facilitate research on understanding the interplay between genes and environmental factors on disease etiology. Data are collected regarding environmental factors, family and lifestyle, clinical experimental outcomes and imaging results of pregnant women and children from birth to 18 years old. Biological samples including blood and tissue samples are also collected from the children and their parents.

DETAILED DESCRIPTION:
Early life phase (fetal and infant) is a critical period for the development of health and disease in a person's life. Many adult chronic diseases, such as diabetes, cardiovascular and cerebrovascular diseases, all come from the exposure of negative environmental and behavioral factors during this period. By collecting the lifestyle data and clinical data of pregnant women at different periods, the appropriate indicators are anticipated to be selected to predict and evaluate the outcome of pregnancy and the health of the mothers and children in the long term. The status of overweight and obesity of children in Shenyang and its surrounding areas are anticipated to be analyzed by descriptive and etiological analysis through collecting the lifestyle data and clinical data of different periods of pregnant women and the lifestyle data of different developmental stages of children.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women, <13 gestational weeks
2. Permanent residents or families intended to remain in Shenyang and surrounding areas
3. Pregnant women who are planned to be examined and delivered in Shengjing Hospital.

Exclusion Criteria:

1. Pregnant women who refuse to take part in the study
2. Pregnant women have diseases that might affect the results of researches, including neuropsychiatric disorders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women in Shenyang, China and their husband and children
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2037-06 (Estimated)

PRIMARY OUTCOMES:
Change of biometric parameter in centimeter of fetuses at the thirteenth week of gestational age | At every week from the thirteenth week of gestational age to delivery of babies
  Including head circumference, abdominal circumference, biparietal diameter, femur length of singleton and twin pregnancy
Weight in kilogram of neonate | At birth of neonate
  Including singleton and twin pregnancy measured by nurses
Gene expression of husbands of pregnancy women | At 13 weeks of gestational age
  DNA methylation, histone acetylation etc. assessed by analyses of blood
Change of gene expression of pregnancy women | At 13, 26 and 34 weeks of gestational age
  DNA methylation, histone acetylation etc. assessed by analyses of blood
Result of Non-invasive Prenatal Testing | From 12 to 22 weeks of gestational age
  including singleton and twin pregnancy

SECONDARY OUTCOMES:
Change of intestinal flora during early childhood | Age at 1 year, 3 years, 6 years, 9 years, 12 years, 15 years and 18 years
  Assessed by analyses of stool samples
Height in centimeter changes during childhood | Age at 1 year, 3 years, 6 years, 9 years, 12 years, 15 years and 18 years
  Measured by nurses in clinic
Weight in kilogram changes during childhood | Age at 1 year, 3 years, 6 years, 9 years, 12 years, 15 years and 18 years
  Measured by nurses in clinic
Change of gene expression during childhood | Age at 1 year, 3 years, 6 years, 9 years, 12 years, 15 years and 18 years
  DNA methylation, histone acetylation etc. assessed by analyses of blood

CONTACTS AND LOCATIONS:
Overall Officials: Caixia Liu, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang L, Du Y, Zhou J, Liu C, Li J, Qiao C. Timing of diagnostic workups in Chinese population with recurrent pregnancy loss: a cross-sectional study. BMC Pregnancy Childbirth. 2025 Mar 29;25(1):373. doi: 10.1186/s12884-025-07330-8. PMID 40158174